CLINICAL TRIAL: NCT00353977
Title: A Pilot Trial of an Accelerated Immunization Schedule With ALVAC-pp65 (vCP260) for Inducing CMV-Specific Immunity in Stem Cell Allotransplant Donors and Healthy Volunteers
Brief Title: Accelerated Immunization to Induce Cytomegalovirus Immunity in Stem Cell Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Minoo Battiwalla, M.D., Principal Investigator, National Heart, Lung, and Blood Institute (NHLBI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 040198; 04-H-0198 (Other: National Heart Lung and Blood Institute)
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-06

CONDITIONS: Cytomegalovirus Infections
Keywords: Cytomegalovirus; Vaccine; CMV; Immunization; Peripheral Blood Stem Cell Transplantation; Stem Cell Allotransplant
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALVAC-CMV (vCP260) Vaccinated group (Experimental): Patients who were vaccinated with ALVAC-CMV (vCP260)
  Interventions: Biological: ALVAC-CMV (vCP260)

INTERVENTIONS:
Biological: ALVAC-CMV (vCP260) — ALVAC-pp65 (vCP260), an attenuated canary pox-based vaccine (Aventis Sanofi Pasteur, Lyon, France), 3 doses (1.0 ml each) delivered intramuscularly in the deltoid muscle.
  Sero-negative subjects will receive a total of 3 immunizations to be given day 0, 5 and 10.
  Sero-positive subjects will receive a total of 2 immunizations to be given day 0 and 5. (Protocol amendment after findings from the 9/6/2006 interim analysis demonstrated that in the sero-positive group, only 2 vaccinations were required to generate maximum immune response.)
  Other Names: Canary Pox CMV vaccine

SUMMARY:
This study will evaluate the safety and effectiveness of a new vaccine, ALVAC-pp65, in boosting immunity to cytomegalovirus (CMV) infection in stem cell transplant donors. CMV is a member of the herpesvirus group, which includes herpes simplex virus types 1 and 2, varicella-zoster virus (which causes chickenpox), and Epstein-Barr virus (which causes infectious mononucleosis). Most adults are infected with CMV, but a healthy immune system keeps the virus in check, so that it does not cause harm. In people with a weakened immune system, such as transplant recipients, the virus can become reactivated. Medications for treating the infection may cause low blood counts and kidney damage, and, in some cases, the virus may cause death. The ALVAC-pp65 vaccine is intended to improve immunity against CMV in stem cell donors and thereby prevent its reactivation in recipients. It is made from a virus that ordinarily infects canaries. The virus is weakened so that it cannot infect the person who receives it, and it is modified to carry a copy of a CMV gene called pp65. This gene instructs cells to make CMV proteins that the vaccine recipient's immune system can produce antibodies to, thus conferring immunity to the disease.

Persons 18 years of age or older who are scheduled to donate stem cells for a patient in an NIH protocol and who are not allergic to eggs, egg products, or other vaccines, may be eligible for this study. Candidates are screened with a medical history, physical examination, and blood tests.

Participants receive three vaccinations one week apart beginning at least 3 weeks before the scheduled stem cell donation. They are observed for 30 minutes after each vaccination to look for any immediate side effects of the vaccine. Approximately 3 tablespoons of blood are drawn before each vaccination and 1 week after the last vaccination to evaluate vaccine safety. Blood samples are also collected at the screening evaluation, 3 weeks after the start of vaccination, and 3 months after the last vaccination to check for CMV immunity.

Participants keep a diary, recording any reactions to the vaccine and any change in medications. They are contacted by telephone for follow-up 3 months after the last vaccination to report any additional symptoms.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) infection is a major complication following allogeneic stem cell transplantation (SCT). The risk of CMV infection after SCT is inversely related to the number of CMV-specific cytotoxic T-lymphocytes (CTLs) present in the allograft. CMV-specific lymphocytes can be readily detected and quantified in the blood by sensitive in vitro techniques that measure T cell cytokine secretion following antigen stimulation. A previous phase I clinical trial has demonstrated that CMV-specific T cells can be safely generated in normal CMV-seronegative (naive) subjects after immunization with the CMV vaccine, ALVAC-pp65 (vCP260), an attenuated canary pox-based vaccine Sanofi Pasteur (formerly known as Aventis Pasteur, Lyon, France).

We propose a clinical trial to evaluate an accelerated immunization schedule with the same vaccine. Study participants will be 1) SCT donors and their matched recipients participating in intramural NIH allogeneic SCT protocols and 2) CMV sero-negative normal volunteers. Donors will receive two or three immunizations prior to allograft collection, and followed for 45 days for the development of CMV immunity. Normal volunteers will receive two or three immunizations and followed similarly to the donors. CMV sero-positive subjects will receive two immunizations; CMV sero-negative subjects will receive three. Transplant (SCT) recipients will be evaluated for incidence of CMV infection and disease.

The study is designed as a two-stage phase II trial with stopping rules at each stage. The primary outcome measures are the effectiveness of the vaccine in (a) generating cellular immunity in CMV-seronegative (naive) donors or CMV sero-negative normal volunteers and (b) boosting the cellular immune response in CMV-seropositive (sensitized) donors and healthy volunteers. Secondary outcomes include the clinical safety profile of the vaccine in vaccine recipients and the incidence of CMV infection/disease in transplant recipients. Since the cellular immune response to CMV is a standard model for immune reconstitution post transplant, our study may also provide important information on the feasibility of immunizing stem cell transplant donors with other microbial and tumor vaccines.

ELIGIBILITY:
- INCLUSION CRITERIA: VACCINE RECIPIENT

* Under evaluation for enrollment as a donor on a stem cell transplant protocol at the NIH Clinical Center, Or
* CMV sero-negative or sero-positive healthy volunteer
* Age greater than or equal to 18 years, but less than or equal to 80 years
* Ability to comprehend the investigational nature of the study and provide informed consent
* All subjects (men and women) must agree to practice abstinence or effective contraception during the study period
* Baseline laboratory evaluations are within normal limits
* For woman, negative urinary pregnancy test
* Informed consent from transplant recipients obtained
* INCLUSION CRITERIA:

STEM CELL TRANSPLANT RECIPIENT

* Under evaluation for enrollment as a recipient on a stem cell transplant protocol at the NIH
* Age greater than or equal to 18 years, and less than or equal to 75 years
* Ability to comprehend the investigational nature of the study and provide informed consent
* EXCLUSION CRITERIA:

VACCINE RECIPIENT

* History of severe adverse reaction or allergy to any vaccine
* Known or suspected allergies to vaccine constituents - eggs, mono-sodium glutamate or neomycin
* Acute febrile illness within the 72 hours preceding the vaccination
* History of any immunosuppressive disease or major chronic disorder
* History of treatment with immunosuppressive medications in the past 6 months
* Pregnant or breast feeding
* Enrolled or planning to enroll in another drug or vaccine clinical trial during the study period (other than the stem cell transplant when applicable)
* EXCLUSION CRITERIA:

STEM CELL TRANSPLANT RECIPIENT

- There are no exclusion criteria for stem cell transplant recipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minocher Battiwalla, MD, Principal Investigator — National Institutes of Health- NHLBI
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gerberding JL. Incidence and prevalence of human immunodeficiency virus, hepatitis B virus, hepatitis C virus, and cytomegalovirus among health care personnel at risk for blood exposure: final report from a longitudinal study. J Infect Dis. 1994 Dec;170(6):1410-7. doi: 10.1093/infdis/170.6.1410. PMID 7995979
- [Background] Bevan IS, Daw RA, Day PJ, Ala FA, Walker MR. Polymerase chain reaction for detection of human cytomegalovirus infection in a blood donor population. Br J Haematol. 1991 May;78(1):94-9. doi: 10.1111/j.1365-2141.1991.tb04388.x. PMID 1645986
- [Background] Bolovan-Fritts CA, Mocarski ES, Wiedeman JA. Peripheral blood CD14(+) cells from healthy subjects carry a circular conformation of latent cytomegalovirus genome. Blood. 1999 Jan 1;93(1):394-8. PMID 9864186
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2004-H-0198.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hematopoietic stem cell transplant (sibling) donors and normal volunteers at a quaternary hospital.
  Recruitment: 3/05 to 11/06
Groups:
- Alvac pp65 Vaccine: Subjects received 2 or 3 doses of the vaccine
Period: Overall Study
Arm/Group | Alvac pp65 Vaccine
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alvac pp65 Vaccine
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Cellular Immune Response in Vaccine Recipients
Description: Evaluate the efficacy of an accelerated ALVAC-pp65 immunization schedule in generating cytomegalovirus (CMV)-specific immunity in seronegative transplant donors and healthy volunteers (HV) and augmenting CMV-specific immunity in seropositive transplant donors.
Time Frame: Day 45
Population: 11 subjects were CMV seropositive and 3 subjects were seronegative.
Measure: Number; unit: participants
Arm/Group | Alvac pp65 Vaccine
Number analyzed (Participants) | 14
participants | 14

ADVERSE EVENTS:
Groups:
- Alvac pp65 Vaccine: Subjects received 1, 2 or 3 doses of the vaccine
Arm/Group | Alvac pp65 Vaccine
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 14/38
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvac pp65 Vaccine (N=38)
hypotension (Cardiac disorders) | 1 (1)
chills (General disorders) | 1 (1)
diaphoresis (General disorders) | 1 (1)
fatigue (General disorders) | 5 (5)
malaise (General disorders) | 3 (3)
rigors (General disorders) | 1 (1)
weakness (General disorders) | 2 (2)
nausea (General disorders) | 1 (1)
swollen lymph nodes, axillary (Blood and lymphatic system disorders) | 4 (4)
dizziness (Nervous system disorders) | 2 (2)
tingling, fingers (Nervous system disorders) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
myalgia (General disorders) | 2 (2)
headache (Nervous system disorders) | 8 (8)
fever (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes